CLINICAL TRIAL: NCT03387202
Title: Uterine Preserving Apical Prolapse Correction With Laparoscopic Lateral Mesh Suspension: Initial Experience by Defining Anatomic and Subjective Success
Brief Title: Laparoscopic Lateral Mesh Suspension for Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, MURAT YASSA, Principal Investigator, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: FSM KAEHK
Record Dates: First submitted 2017-04-01; First posted 2018-01-02 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Pelvic Organ Prolapse; Pelvic Floor Prolapse
Keywords: Pelvic Organ Prolapse; Translabial ultrasound; Transperineal ultrasound; Lateral Mesh Suspension; Descensus uteri; Laparoscopic pelvic organ prolapse repair
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pelvic organ prolapse: Participants received "Laparoscopic lateral suspension with mesh" as part of routine medical care in apical prolapse, thus, the investigator does not assign a intervention but studies the effects.Vaginal length, bladder neck mobility and pelvic floor biometry with AP hiatal diameter and pelvic organ descent measurements are measured by Transperineal ultrasound to assess anatomic success in the preoperative and at postoperative 18th months. POP-Q assessment and translabial usg for objective success; Female Sexual Function Index (FSFI), Michigan Incontinence Severity Index (M-ISI), Prolapse Quality of Life questionnaire (PQoL), Pelvic Organ Prolapse Symptom Score (POP-SS) and Visual Analog Score (VAS) are used to assess subjective success.
  Interventions: Procedure: Laparoscopic lateral suspension with mesh; Diagnostic Test: Transperineal ultrasound

INTERVENTIONS:
Procedure: Laparoscopic lateral suspension with mesh — V-shaped ccm wide and 25cm length mesh strip is prepared from a 30x30cm Prolene mesh (Ethicon J&J).Deep dissection of the uterovesical space is performed.Cutaneous incisions are bilaterally made 3cmsuperoposterior to the anteriosuperior iliac spine.A grasper is introduced retroperitoneally through the subperitoneum holding the beginning part of mesh until reaching the vesicovaginal space in an oblique route rather than transverse.Broad ligament is lifted upward and tunnel is practiced in its lower third.Assistant grasper catches the distal mesh and pulls out through the opposite subperitoneal tunnel.Corner of mesh is fixed to the pubocervical fascia,uterine cervix and isthmus with Absorba Tack™(Covidien, Mansfield,USA).Tension-free lateral mesh suspension is achieved at the desired level
Diagnostic Test: Transperineal ultrasound — Vaginal length, bladder neck mobility and pelvic floor biometry with anterioposterior hiatal diameter and pelvic organ descent measurements are measured by transperineal ultrasonography to assess anatomic success in the preoperative and at postoperative first third and sixth months if available.
  Other Names: Translabial ultrasound

SUMMARY:
This study is aimed to share our clinical experience in an uterine-preserving laparoscopic lateral suspension of apical prolapses with mesh operation after minor modifications in technique. Transperineal ultrasonography and several questionnaires are used for objective and subjective outcomes.

DETAILED DESCRIPTION:
Vaginal length, bladder neck mobility and pelvic floor biometry with anteroposterior hiatal diameter and pelvic organ descent measurements are measured by transperineal ultrasonography to assess anatomic success in the preoperative and at postoperative 18th months if available.

Female Sexual Function Index (FSFI), Michigan Incontinence Severity Index (M-ISI), Prolapse Quality of Life questionnaire (PQoL), Pelvic Organ Prolapse Symptom Score (POP-SS) and Visual Analog Score (VAS) are used to assess subjective success in the preoperative and at postoperative 18th months if available.

,

ELIGIBILITY:
Inclusion Criteria:

* >18 years old symptomatic women with pelvic organ prolapse needing surgery.
* Patients who are not comfortable with using or refusing pessary
* Refusing sacrocolpopexy due to its serious surgical risk

Exclusion Criteria:

* Patients who prefer sacrocolpopexy
* Any cue for gynecologic oncological condition
* Patients who approves Le Fort colpocleisis among who does not have any sexual intercourse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic women with pelvic organ prolapse
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline POP-Q measurements (mm) at 18th month. | 18 months
  Prolapse degree; Point Ba/C/Bp

SECONDARY OUTCOMES:
Subjective Success - Change from baseline Female Sexual Function Index (FSFI) to measure sexual dysfunction at 18th month. | 18 months
  Validated into Turkish language form will be used to compare preoperative and postoperative period. The FSFI is a multiple-trait scoring, self-report document used to assess female SF during the previous 4 weeks. It consists of 19 items that encompass six separate domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. The maximum score is 36 points and the minimum score is 2 points. After completion of the questionnaire, the total SF score was calculated as follows: no sexual dysfunction (SD) (≥ 30 points) , mild SD (between <29 and > 23 points), and severe SD (≤ 22 points).
Subjective Success - Change from baseline Michigan Incontinence Severity Index (M-ISI) to measure urinary incontinence at 18th month. | 18 months
  Validated into Turkish language form will be used to compare preoperative and postoperative period. It has ten items, consisting of a total M-ISI domain (the sum of items 1-8) and a distinct Bother domain (the sum of items 9 and 10). The total M-ISI score consists of three subdomains (items 1-3 for stress urinary incontinence [SUI], items 4-6 for UUI, and items 7 and 8 for PU). The responses for each item range from 0 to 4 on a Likert-type scale, with higher values representing greater symptoms and greater bother. The total M-ISI domain ranges from 0 to 32, the Bother domain ranges from 0 to 8, the SUI and UUI subdomains range from 0 to 12, and the PU subdomain ranges from 0 to 8. Total domain and subdomain scores are obtained by simply adding the respective answers. The minimally important difference has been determined for the following domains/subdomains: total M-ISI (4 points), SUI (2 points), UUI (2 points), and PU (1 point).
Subjective Success - Change from baseline Prolapse Quality of Life questionnaire (PQoL) to measure quality of life according to pelvic organ prolapse at 18th month. | 18 months
  Validated into Turkish language form will be used to compare preoperative and postoperative period. he questionnaire included 20 questions grouped in sections (domains) related to a particular aspect of quality of life. A total of nine domains covering general health, prolapse impact, role limitations, physical and social limitations, personal relationships, emotional problems, sleep/energy disturbance as well as severity symptoms measurements were defined. Questions regarding bladder, bowel and sexual function were also separately included and validated for reproducibility and internal consistency. Responses ranged from 'none/not at all', through 'slightly/a little' and 'moderately' to 'a lot' to produce a four-point scoring system for each item. Scores in each domain ranged between 0 and 100 with a high total score indicating a greater impairment of quality of life.
Subjective Success - Change from baseline Pelvic Organ Prolapse Symptom Score (POP-SS) to measure quality of life according to pelvic organ prolapse at 18th month. | 18 months
  Validated into Turkish language form will be used to compare preoperative and postoperative period. Total range scores: 28 (min:0, max:28). Higher values represent a worse outcome.
Subjective Success - Change from baseline Visual Analog Score (VAS) for pain at 18th month. | 18 months
  Participant describes the pain related to the mesh. The respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain with a format of a horizontal bar.
Change from baseline Pelvic Hiatus measurements (mm) at 18th month. | 18 months
  Anteroposterior hiatal length (mm)
Change from baseline Pelvic biometry measurements at 18th month. | 18 months
  Prolapse degree over symphysis pubis (mm) Anterior compartment over 10, Posterior compartment over 15 mm are clinically relevant
Change from baseline bladder neck mobility measurements at 18th month. | 18 months
  Urethral rotation (degree) between rest and valsalva maneuver states
Failure (%) | 18 months
  Failure is defined by any recurrence of prolapse, mesh erosion and need for additional surgery

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol
Time Frame: Immediately, until the publishing
Access Criteria: Study protocol can be sent upon request murat.yassa@gmail.com